CLINICAL TRIAL: NCT06455748
Title: Daratumumab/Daratumumab and Hyaluronidase-fihj in Combination With Pomalidomide and Dexamethasone for the Treatment of Patients With Newly Diagnosed AL Amyloidosis: a Prospective, Multicenter, Single-arm Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yongyong MA (Other)
Responsible Party: Sponsor-Investigator, Yongyong MA, Chief Physician of Hematology Department, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Poma-DD-AL-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Amyloid Light-chain Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; darlin protein, Dictyostelium; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab/daratumumab and hyaluronidase-fihj in combination with pomalidomide, dexamethasone (DPd) (Experimental): Observed patients meeting the screening criteria were treated with Daratumumab/daratumumab and hyaluronidase-fihj + pomalidomide + dexamethasone regimen as appropriate.
  Combined regimen of the above until disease progression or up to 2 years.
  Interventions: Drug: Daratumumab/daratumumab and hyaluronidase-fihj; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab/daratumumab and hyaluronidase-fihj — Daratumumab/daratumumab and hyaluronidase-fihj: Dara SC 1800mg subcutaneous (IH) or Dara 16mg/kg intravenously (IV) administered weekly (qwk) x 4 every 2 weeks X 3 doses per month starting C7.
  Other Names: Dara
Drug: Pomalidomide — Pomalidomide: pom 2-4mg PO day (D) 1-21/28 (adjust dose for renal function).
  Other Names: pom
Drug: Dexamethasone — Dexamethasone: dex C1: 20mg IV D1/8, 20mg PO D2/9 and 40mg PO C1D15 weekly up to C6, then 20mg IV monthly starting C7D1 and 20mg PO D8, 15, 22.
  Other Names: dex

SUMMARY:
This is a prospective and single arm clinical study. The goal of this clinical trial is to observe and evaluate the efficacy and safety of Daratumumab/daratumumab and hyaluronidase-fihj in combination with pomalidomide and dexamethasone in the treatment of patients with newly diagnosed AL amyloidosis.

DETAILED DESCRIPTION:
Primary objective:

Hematologic overall remission rate (ORR) as defined by the criteria in the Chinese Guidelines for the Diagnosis and Treatment of Systemic Light Chain Amyloidosis, 2021 edition.

Secondary objective:

1. organ remission rate as defined by the criteria of the Chinese Guidelines for the Diagnosis and Treatment of Systemic Light-Chain Amyloidosis 2021 Edition, hematologic complete remission (CR) rate, very good partial remission (VGPR) rate, progression free survival (PFS), overall survival (OS), and negative rate of microscopic residual disease (MRD).
2. safety of combination therapy regimens.

Exploratory purpose:

EORTC QLQ-C30.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, diagnosed with primary amyloidosis of AL tissue;
2. ECOG PS score 0-2 points;
3. Measurable disease: The difference between affected and unaffected FLC is>20 mg/L, and the serum immunoglobulin kappa λ FLC ratio is abnormal;
4. Having sufficient organ and bone marrow function, defined as follows:

   1. Blood routine: Absolute neutrophil count ≥ 1.0 x 10 ^ 9/L, platelet count ≥ 50 x 10 ^ 9/L;
   2. Blood biochemistry and electrolytes: ALT and AST both ≤ 3 times the upper limit of normal, total bilirubin ≤ 1.5 times the upper limit of normal, creatinine clearance rate ≥ 30 mL/min, serum corrected calcium ≤ 14.0 mg/dL (≤ 3.5 mmol/L) or free ion calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L);
5. Women of childbearing age must agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 3 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test was negative and must be a non lactating patient; In addition, if the subject misses their menstrual period or experiences abnormal menstrual bleeding, the researcher can conduct a pregnancy trial at any time during the study period;
6. Men must agree to use contraceptive measures during the study period and within 3 months after the end of the study period;
7. The patient agrees to participate in the clinical trial and signs an informed consent form.

Exclusion Criteria:

1. Non AL amyloidosis;
2. Known to be allergic, hypersensitive or intolerant to monoclonal antibodies or human derived proteins, daretozumab or its excipients, or known to be allergic to mammalian derivatives;
3. Female patients who have tested positive for lactation or serum pregnancy test during the screening period;
4. Received ASCT or had graft-versus-host disease in the past 12 months;
5. Suffering from moderate or severe persistent asthma within 2 years prior to enrollment, or having uncontrolled asthma at the time of enrollment;
6. Evidence of having other malignant tumors within the 3 years prior to enrollment or having been previously diagnosed with another malignant tumor with any residual lesions;
7. Suffering from chronic obstructive pulmonary disease (COPD), the forced expiratory volume (FEV1) in one second is less than 50% of the normal expected value;
8. Clinically significant heart disease, including:

   1. Start studying myocardial infarction or unstable or uncontrollable conditions within 6 months prior to treatment (such as unstable angina, congestive heart failure, New York Heart Association (NYHA) III-IV);
   2. Arrhythmias (NCI CTCAE V5.0 standard ≥ grade 3) or clinically significant electrocardiogram (ECG) abnormalities;
   3. The electrocardiogram shows a baseline corrected QT (QTc) interval>470 ms;
9. Active infections, including but not limited to HAV, HBV, HCV, HIV;
10. Plasma cell leukemia (circulating plasma cells>2.0 × 10 ^ 9/L) or Waldenstrom macroglobulinemia (WM) or POEMS syndrome (multiple neuropathies, organ enlargement, endocrine disorders, monoclonal plasma cell disease, and skin changes);
11. Peripheral neuropathy or neuralgia of grade 2 or above (CTCAE 5.0 standard);
12. Underwent major surgery within 14 days prior to enrollment, or did not fully recover from early surgery, or planned surgery during the study period or within 14 days after the last study drug treatment (note: does not include surgery under local anesthesia or kyphoplasty or vertebroplasty);
13. According to the judgment of the investigator, there are concomitant diseases (such as active systemic infection, uncontrolled diabetes, acute diffuse invasive pulmonary disease, neurological or mental disease, etc.) or any other conditions that may confuse the research results or affect the completion of the study;
14. Individuals who are receiving any other experimental drugs or experimental medical devices;
15. The researchers believe that the patient has other circumstances that are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Hematologic Overall Remission Rate (ORR) | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  ORR was defined as the proportion of subjects who achieved partial remission (PR) or better partial remission (VGPR) and complete response (CR) by Guideline 2021 Edition criteria.

SECONDARY OUTCOMES:
Hematologic complete remission (CR) rate | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  Negative blood/urine immunofixation electrophoresis and normal serum free light chain levels and ratios.
Very good partial remission (VGPR) rate | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  dFLC decreased to <40 mg/L
Overall survival (OS) | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  OS: defined as the time from the start of the subject's randomization enrollment until death or final follow-up (time lost to follow-up).
Progression free survival （PFS） | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  PFS was defined as the period from the subject's randomization to enrollment to the date of the first documented disease progression (PD) (rated according to IMWG criteria, with or without continuation of treatment) or the date of death from any cause, whichever occurred first.
Negative rate of microscopic residual disease (MRD) | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  MRD level: MRD was detected using second-generation sequencing (NGS) for bone marrow MRD levels. MRD negative rate: MRD is only evaluated in patients who achieve CR or better.
Time to response (TTR) | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  TTR: defined as the period from randomization of subjects to the date of first recorded disease remission.
Duration of response (DOR) | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  DOR: defined as the date from the first recording of treatment response to the first recording of disease progression or the date of death from any cause.

OTHER OUTCOMES:
Adverse event | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  An adverse event is defined as an adverse medical event that occurs after a patient in a clinical trial has received treatment in this study, but is not necessarily causally related to the treatment. Any adverse medical event that occurred in this trial from the time the patient signed the informed consent form until 30 days after the final treatment was determined to be an adverse event, regardless of whether it was causally related to the study treatment.
EORTC QLQ-C30 | A follow-up is required 30 days (± 7 days) after the completion of all treatments, followed by a follow-up every 12 weeks (± 7 days) for a period of 1 year.
  EORTC QLQ-C30 is the core scale developed by the European Organization for Research and Treatment (EORTC) for measuring the quality of life of cancer patients. It is used for measuring the common components of quality of life in all cancer patients, and on this basis, specific items (modules) for different cancers are added to form specific scales for different cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Yongyong Ma, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No